CLINICAL TRIAL: NCT04187885
Title: Effect of Physical Activity Program During Academic Stress on Adolescent Sleep
Brief Title: Physical Activity Stress and Sleep in Adolescents
Acronym: APADOSLEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose (Other)
Collaborators: Biochimie Clinique LR99ES11 (Unknown); Department of Biochemistry, La Rabta Hospital, Tunisia. (Unknown); Université de Toulon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: University Tunis El Manar
Record Dates: First submitted 2019-09-20; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Adolescent Problem Behavior
Keywords: sleep; adolescent; physical activity; academic stress
MeSH Terms: conditions — Motor Activity | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group/Cohort 1 : CTL (Active Comparator): Label : control
  Type : comparator
  Description: Outside academic stress period (represented by exams), without the physical activity program (no Intervention).
  Interventions: Behavioral: Group/Cohort 2: PAP
- Group/Cohort 2: PAP (Experimental): Label : physical activity program without stress Type : experimental
  Description: outside academic stress period (exams), with the physical activity program:60 min of mederate to vigorous leisure activities and exercises will be proposed from Monday to Thursday.
  Interventions: Behavioral: Group/Cohort 2: PAP
- Group/Cohort 3: AS (Experimental): Label : academic stress Type : experimental
  Description: during academic stress period (exams), without the physical activity program (no Intervention)
  Interventions: Behavioral: Group/Cohort 2: PAP
- Group/Cohort 4: ASPAP (Experimental): Label : academic stress and physical activity program Type : experimental Description: during academic stress period (exams), with the physical activity program: 60 min of mederate to vigorous leisure activities and exercises will be proposed from Monday to Thursday.
  Interventions: Behavioral: Group/Cohort 2: PAP

INTERVENTIONS:
Behavioral: Group/Cohort 2: PAP — Each experimental session will be carried out over 5 days of a week. Adolescents will take part randomly in four sessions.
  Physical activity program will be identical between sessions and groups. 60 min of moderate to vigorous leisure activities and exercises will be proposed each day. Heart rate monitor will be used to control intensity of exercise during the physical activity program.
  Other Names: Physial activity Program

SUMMARY:
Adolescence is characterized by major transitions in sleep and circadian rhythm. This rapid pivotal period increases the risks of sleep debt and poor sleep quality, leading to pronounced diurnal fatigue and drowsiness. On the other hand, academic stress has been also associated with increased sleep disturbances.

Both academic stress and poor sleep in adolescents has been linked to increased sleepiness rate, reduced alertness, lower academic performances and the impairment of the control of energy balance through hyperphagia.

Despite the importance of sleep in holistic development, physical (i.e. recovery, metabolism, muscle growth, weight control), cognitive (i.e. learning, memory, decision-making, Vigilance). Few studies have been designed to improve this behavior among college adolescents, especially in times of academic stress.

Physical activity has been suggested as a non-pharmacological alternative treatment for sleep disorders . Generally, it is well established that the duration and quality of sleep were improved by regular physical activity among adolescents and far better, it was suggested that the exercise-mediated effect on sleep could be even observed in the short term. Moreover, it was suggested that aerobic exercise has positive effects on psychological stress and well-being of adolescents .

Therefore, APADOSLEEP trial, was designed to examine the effect of physical activity program on sleep during and outside periods of academic stress.

DETAILED DESCRIPTION:
Counterbalanced, cross-over, pre-post trial where each subject acts as his own control.

Four sessions will be performed for each adolescent. Each session will be conducted over 5 days (from Monday to Friday):

Adolescents will take part randomly in four sessions. Physical activity program will be identical between sessions and groups. 60 minn of moderate to vigorous leisure activities and exercises will be proposed each day. Heart rate monitor will be used to control intensity of exercise during the physical activity program.

* Control session (CTL) outside academic stress period (represented by exams) and without the physical activity program.
* A session outside academic stress period, with the physical activity program (PAP).
* A session during an academic stress period without the physical activity program (AS).
* A session during an academic stress period with the physical activity program (ASPAP).

At each session:

* Continuous sleep assessments (duration and quality) by accelerometry
* Continuous physical activity and sedentary behaviour assessments by accelerometry
* one evaluation of melatonin peak from salivary specimens
* one evaluation of cortisol peak from salivary specimens
* An evaluation of the ad libitum food intake of the 5th day will be carried out by the weighing method.
* one assessment of cognitive performance
* An evaluation of subjective appetite sensations (hunger, fullness, desire to eat) of the 5th day
* An evaluation of subjective diurnal sleepiness (Karolinska) of the 5th day

ELIGIBILITY:
Inclusion Criteria:

* college adolescent Tanner stages 3-5

Exclusion Criteria:

* Disorders and / or pathology of sleep
* Medical or surgical history not compatible with the study, any other chronic illness or injury that may interfere with the subject's abilities
* Take medication that may interfere with the results of the study (corticosteroids ...) or sleeping pills
* Surgical intervention in the previous 3 months
* Regular consumption of tobacco, cannabis or alcohol
* Special diet

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2020-09-03 (Estimated); Primary Completion 2021-11-28 (Estimated); Study Completion 2022-03-03 (Estimated)

PRIMARY OUTCOMES:
sleep Efficiency (%) | change from baseline at 4th night
  the percentage of time spent asleep while in bed

SECONDARY OUTCOMES:
bedtime | change from baseline at 4th night
  the time when the subjet goes to bed
total time in bed (minutes) | change from baseline at 4th night
  total time spent in bed
sleep onset latency (minutes) | change from baseline at 4th night
  actual time it takes to transition from wake to sleep in minutes
wake after sleep onset | change from baseline at 4th night
  awke after sleep has been initiated and before final awake
nubmer of awake >3 minutes | change from baseline at 4th night
  awkenings >3 minutes after sleep has been initiated and before final awake
Sedentary activities | pre and post intervention:day 1 and day 4
  time spent on Sedentary activities < 1Metabolic Equivalent of task (METs),
light activities | pre and post intervention:day 1 and day 4
  time spent on [1 - 3 ] expressed in Metabolic equivalent of task (METs)
moderate to vigorous activities | pre and post intervention : day1 and day 4
  time spent on moderate to vigorous activities [3 - 9 Metabolic equivalent of task[
Energy expenditure (kilo calories) | pre and post intervention : day1 and day 4
  the amount of energy a person uses in the form of calories estimated by accelerometers
circadian phase (DLMO) | night 4
  evaluations of melatonin peak from salivary specimens (5 measures), time (180, 120, 60 min before bedtime, bedtime and 60 min after bedtime)
Cortisol peak | day 5
  evaluations of cortisol peak from salivary specimens (5 measures), (upon awakening, awakening + 30mn, awakening + 60mn, awakening + 120mn et awakening + 180mn)
Stroop test | day 5
  selective attention and reading ability
Trail marking test | day 5
  this test estimate visual attention and motor speed
Barrage test | day 5
  this task evaluates visual- spatial ability and recognition
California verbal learning test. | day 5
  this test evaluates primary and secondary memory
Energy intake | day 5
  Energy intake and proportion of the energy derived from each class of macronutrients (carbohydrate, fat, and protein) measured on meals offered "ad-libitum"
Subjective appetite sensations | day 5
  hunger, fullness, desire to eat and prospective food consumption : upon awakening, before and right after the breakfast, lunch, snack and dinner as well as bed time.
  Appetite sensations will be collected throughout the day using visual analogue scales (150 mm scales). Adolescents will report their hunger, fullness, desire to eat and prospective food consumption at thirteen regulated times: upon awakening, before and right after the breakfast, lunch, snack and dinner as well as bed time. The questions were i) "How hungry do you feel?", ii) "How full do you feel?", iii) "Would you like to eat something?", iv) "How much do you think you can eat?" (adolescents were asked to respond on a scale from "not at all" to "a lot"). This method has been previously validated
Subjective sleepiness (Karolinska scale) | day 5
  this scale mesures the subjective level os sleepness at particular times during the day. this is a nine point scale (1= extreemly alert, 3= alert, 5= neither nor sleepy, 7 = sleepy but no difficulty for main awake, 9= extreemly sleepy/ fighting sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Amani Kallel, PHD, Principal Investigator — Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora, T., and Grey, I. (2019). Sleep, obesity and cardiometabolic disease in children and adolescents. In Sleep and Health, (Elsevier), pp. 421-433.
- [Background] Colrain IM, Baker FC. Changes in sleep as a function of adolescent development. Neuropsychol Rev. 2011 Mar;21(1):5-21. doi: 10.1007/s11065-010-9155-5. Epub 2011 Jan 12. PMID 21225346
- [Background] Dewald JF, Meijer AM, Oort FJ, Kerkhof GA, Bogels SM. The influence of sleep quality, sleep duration and sleepiness on school performance in children and adolescents: A meta-analytic review. Sleep Med Rev. 2010 Jun;14(3):179-89. doi: 10.1016/j.smrv.2009.10.004. Epub 2010 Jan 21. PMID 20093054
- [Background] Haugland S, Wold B, Torsheim T. Relieving the pressure? The role of physical activity in the relationship between school-related stress and adolescent health complaints. Res Q Exerc Sport. 2003 Jun;74(2):127-35. doi: 10.1080/02701367.2003.10609074. PMID 12848225
- [Background] Ivanenko A, Crabtree VM, Gozal D. Sleep and depression in children and adolescents. Sleep Med Rev. 2005 Apr;9(2):115-29. doi: 10.1016/j.smrv.2004.09.006. PMID 15737790
- [Background] Kredlow MA, Capozzoli MC, Hearon BA, Calkins AW, Otto MW. The effects of physical activity on sleep: a meta-analytic review. J Behav Med. 2015 Jun;38(3):427-49. doi: 10.1007/s10865-015-9617-6. Epub 2015 Jan 18. PMID 25596964
- [Background] Krietsch KN, Chardon ML, Beebe DW, Janicke DM. Sleep and weight-related factors in youth: A systematic review of recent studies. Sleep Med Rev. 2019 Aug;46:87-96. doi: 10.1016/j.smrv.2019.04.010. Epub 2019 Apr 23. PMID 31100467
- [Background] Lang C, Brand S, Feldmeth AK, Holsboer-Trachsler E, Puhse U, Gerber M. Increased self-reported and objectively assessed physical activity predict sleep quality among adolescents. Physiol Behav. 2013 Aug 15;120:46-53. doi: 10.1016/j.physbeh.2013.07.001. Epub 2013 Jul 9. PMID 23851332
- [Background] Lang C, Kalak N, Brand S, Holsboer-Trachsler E, Puhse U, Gerber M. The relationship between physical activity and sleep from mid adolescence to early adulthood. A systematic review of methodological approaches and meta-analysis. Sleep Med Rev. 2016 Aug;28:32-45. doi: 10.1016/j.smrv.2015.07.004. Epub 2015 Aug 5. PMID 26447947
- [Background] Lund HG, Reider BD, Whiting AB, Prichard JR. Sleep patterns and predictors of disturbed sleep in a large population of college students. J Adolesc Health. 2010 Feb;46(2):124-32. doi: 10.1016/j.jadohealth.2009.06.016. Epub 2009 Aug 3. PMID 20113918
- [Background] Norris R, Carroll D, Cochrane R. The effects of physical activity and exercise training on psychological stress and well-being in an adolescent population. J Psychosom Res. 1992 Jan;36(1):55-65. doi: 10.1016/0022-3999(92)90114-h. PMID 1538350
- [Background] Stepanski EJ, Wyatt JK. Use of sleep hygiene in the treatment of insomnia. Sleep Med Rev. 2003 Jun;7(3):215-25. doi: 10.1053/smrv.2001.0246. PMID 12927121